CLINICAL TRIAL: NCT06443892
Title: Comparison of Postoperative Analgesic Efficacy of Pericapsular Nerve Block (PENG) and Suprainguinal Fascia Iliaca Compartment Block(SFICB) in Intertrochanteric Femur Fractures
Brief Title: Comparison of Pain Relief After Hip Fracture Surgery: Hip and Groin Nerve Block
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: BSH-ANES-MA-01
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Opioid Use; Pain, Postoperative; Hip Fractures
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PENG Group: Participants with intertrochanteric femur fractures undergoing surgery under spinal anesthesia and receiving postoperative pericapsular nerve block (PENG).
  Interventions: Procedure: Pericapsular Nerve Block (PENG)
- SFICB Group: Participants with intertrochanteric femur fractures undergoing surgery under spinal anesthesia and receiving postoperative suprainguinal fascia iliaca compartment block (SFICB).
  Interventions: Procedure: Suprainguinal Fascia Iliaca Compartment Block (SFICB)

INTERVENTIONS:
Procedure: Pericapsular Nerve Block (PENG) — Evaluation of postoperative analgesic efficacy of PENG block in participants with intertrochanteric femur fractures undergoing surgery under spinal anesthesia.
  Groups: PENG Group
Procedure: Suprainguinal Fascia Iliaca Compartment Block (SFICB) — Evaluation of postoperative analgesic efficacy of SFICB block in participants with intertrochanteric femur fractures undergoing surgery under spinal anesthesia.
  Groups: SFICB Group

SUMMARY:
This observational prospective double-blind study aims to compare the analgesic effectiveness of the pericapsular nerve group block (PENG) group and the suprainguinal fascia iliaca compartment block(SFICB) group to be applied to relieve postoperative pain in participants over the age of 18 who will be treated under spinal anesthesia with intertrochanteric femur fracture. The main question it aims to answer is:

* Demonstration of whether PENG block or SFICB is more effective for postoperative analgesia in patients who have undergone intertrochanteric femur fracture surgery, based on pain scores, opioid consumption and patient satisfaction.

ıntertrochanteric femur fractures cause severe pain with movement. Postoperatively, participants' movements are severely restricted, increasing the likelihood of complications.

In this study, participants' pain status, VAS score, opioid consumption through patient-controlled analgesia, and satisfaction will be measured with a survey at the end of the 24th hour.

DETAILED DESCRIPTION:
Intertrochanteric femoral fracture accounts for approximately 45% to 50% of all hip fractures. Intertrochanteric femur fractures cause severe pain with movement. Postoperatively, the movements of the participants are severely restricted, which increases the risk of deep vein thrombosis in the lower extremities, pulmonary infection and mortality in the participants.

Peripheral nerve blocks have been shown to have less impact on hemodynamics, respiratory function, and consciousness than systemic pain relief options. It is recommended as a first-line analgesia program, especially for hip surgeries, with its features of shortening postoperative recovery time, reducing the risk of pneumonia, and not hindering postoperative movement. Fascia Iliaca compartment block used in this area is safe and widely used in postoperative hip fractures. However, to provide effective analgesia for hip surgery, it is necessary to simultaneously block the femoral nerve, lateral femoral cutaneous nerve, and obturator nerve. It has been reported that suprainguinal fascia iliaca compartment block does not provide adequate analgesia and does not reduce opioid consumption because the obturatory nerve cannot be blocked. Therefore, blocking the femoral nerve, obturatory nerve and accessory obturatory nerves with PENG block has led to the idea that postoperative pain scores and opioid consumption will decrease significantly. In this study, we aim to compare the effectiveness of suprainguinal fascia iliaca compartment block and PENG block for postoperative analgesia based on pain scores and opioid consumption in intertrochanteric femur fractures.

Pain is a symptom known to be subjective, and in order to minimize differences between participants, it will be questioned with the Numeric Rating Scale (NRS), which is a standardized scale.

The total narcotic analgesic needs of the block-treated participants will be recorded with the PCA device inserted intravenously postoperatively, and their total Tramadol consumption will be recorded.

Mobilization start times and pain during the mobilization process will be questioned with the Turkish-American Pain Society Revised Patient Outcomes Survey.

The Turkish version of the revised American Pain Society patient outcomes survey for surgical patients will be used to evaluate participants' satisfaction with pain management. According to the confirmatory factor analysis fit indices of the Turkish-Revised American Pain Society Patient Outcomes Questionnaire, whose Cronbach's Alpha value was calculated as 0.88, its three-factor structure was found to be appropriate. The Turkish-Revised American Pain Society Patient Outcomes Questionnaire is a tool to improve the quality of pain management for adult patients. With this questionnaire (1) pain intensity and relief; (2) the impact of pain on activity, sleep, and negative emotions; (3) medication side effects; (4) usefulness of pain management information;(5) ability to participate in pain management decisions; and (6) the use of non-pharmacological techniques will be questioned.

Demographic characteristics of the participants, comorbidities, operation times and complications will be recorded and analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Those with Interthorachanteric Femur Fracture
* Patients over 18 years of age
* ASA I-II-III
* Fully oriented and able to cooperate
* Patients who underwent PENG or Suprainguinal Fascia iliaca compartment block for postoperative analgesia after elective surgery.

Exclusion Criteria:

* ASA IV-V
* Patients under 18 years of age
* Presence of active infection in the area to be treated
* Chronic analgesic use
* Patients who cannot cooperate with postoperative pain follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who underwent surgery under spinal anesthesia with interthorachanteric femur fracture over the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness on pain scores | At 0, 1, 6, 12 and 24 hours after postoperative peripheral nerve block application
  Postoperative pain assessment is performed using the Numerical Rating Scale (NRS). Participants are asked about their rest pain at 0, 1, 6, 12 and 24 hours after applying a postoperative peripheral nerve block. With this method, participants rate their pain with a precise numerical value from 0 to 10. While zero(0) represents "no pain"; Ten (10) represents the opposite end of the pain continuum (e.g., "The most intense pain imaginable," "As intense pain as possible," "Maximum pain").

SECONDARY OUTCOMES:
Effect on total narcotic analgesic consumption | Total number of bolus doses administered at the end of 24 hours of the intravenous PCA device inserted simultaneously after postoperative peripheral nerve block application
  After the surgery, participants will receive a peripheral nerve block procedure in the postoperative anesthetic care area, and then simultaneously receive intravenous patient-controlled analgesia (PCA) and start an infusion. "Tramadol" was preferred as the treatment method to be used for the PCA method. In preparation for PCA, 400 mg of tramadol is added to 100 cc of physiological saline. As PCA protocol, 1 cc/hour (4 mg/hour) basal infusion dose, 5 cc (20 mg) bolus dose, 30 minutes lockout period (maximum 2 bolus doses in 1 hour) are set. The total number of bolus doses administered by the participants on the PCA device at the end of 24 hours will be recorded and evaluated as the amount of additional opioid needed.

OTHER OUTCOMES:
Patient satisfaction | At the end of the patient-controlled analgesia procedure
  The Turkish version of the revised American Pain Society patient outcomes survey for surgical patients will be used to evaluate patients' satisfaction with pain management. According to the confirmatory factor analysis fit indices of the Turkish-Revised American Pain Society Patient Outcomes Questionnaire, whose Cronbach's Alpha value was calculated as 0.88, its three-factor structure was found to be appropriate. The Turkish-Revised American Pain Society Patient Outcomes Questionnaire is a tool to improve the quality of pain management for adult patients. With this questionnaire (1) pain intensity and relief; (2) the impact of pain on activity, sleep, and negative emotions; (3) medication side effects; (4) usefulness of pain management information;(5) ability to participate in pain management decisions; and (6) the use of non-pharmacological techniques will be questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Çam Ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Result] Mosaffa F, Taheri M, Manafi Rasi A, Samadpour H, Memary E, Mirkheshti A. Comparison of pericapsular nerve group (PENG) block with fascia iliaca compartment block (FICB) for pain control in hip fractures: A double-blind prospective randomized controlled clinical trial. Orthop Traumatol Surg Res. 2022 Feb;108(1):103135. doi: 10.1016/j.otsr.2021.103135. Epub 2021 Oct 29. PMID 34715388
- [Result] Kong M, Tang Y, Tong F, Guo H, Zhang XL, Zhou L, Ni H, Wang B, Liu Y, Liu J. The analgesic efficacy of pericapsular nerve group block in patients with intertrochanteric femur fracture: A randomized controlled trial. PLoS One. 2022 Oct 13;17(10):e0275793. doi: 10.1371/journal.pone.0275793. eCollection 2022. PMID 36227845
- [Result] Allard C, Pardo E, de la Jonquiere C, Wyniecki A, Soulier A, Faddoul A, Tsai ES, Bonnet F, Verdonk F. Comparison between femoral block and PENG block in femoral neck fractures: A cohort study. PLoS One. 2021 Jun 4;16(6):e0252716. doi: 10.1371/journal.pone.0252716. eCollection 2021. PMID 34086782
- [Result] Choi YS, Park KK, Lee B, Nam WS, Kim DH. Pericapsular Nerve Group (PENG) Block versus Supra-Inguinal Fascia Iliaca Compartment Block for Total Hip Arthroplasty: A Randomized Clinical Trial. J Pers Med. 2022 Mar 6;12(3):408. doi: 10.3390/jpm12030408. PMID 35330408
- [Result] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544